CLINICAL TRIAL: NCT00380068
Title: ARIES-3: A Phase 3, Long-Term, Open-Label, Multicenter Safety and Efficacy Study of Ambrisentan in Subjects With Pulmonary Hypertension
Brief Title: Safety and Efficacy Study of Ambrisentan in Subjects With Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-323; ARIES-3
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ambrisentan (Experimental)
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Oral tablets taken once daily.
  Other Names: Letairis; Volibris

SUMMARY:
The primary objective of this study was to evaluate the safety and efficacy of ambrisentan in a broad population of participants with pulmonary hypertension (PH). Secondary objectives of this study were to evaluate the effects of ambrisentan on other clinical measures of pulmonary arterial hypertension (PAH), long-term treatment success, and survival.

DETAILED DESCRIPTION:
This study was to enroll up to 200 participants with PH due to the following etiologies: 1) PAH including idiopathic and familial PAH and PAH associated with collagen vascular disease, congenital systemic-to-pulmonary shunts (including Eisenmenger's syndrome), human immunodeficiency virus (HIV) infection, drugs and toxins, thyroid disorders, glycogen storage disease, Gaucher disease, hemoglobinopathies, and splenectomy (WHO Group 1); 2) PH associated with lung diseases and/or hypoxemia, including chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), sleep-disordered breathing, and alveolar hypoventilation disorders (WHO Group 3); 3) PH due to proximal or distal chronic thromboembolic obstruction (WHO Group 4); and 4) PH due to sarcoidosis (WHO Group 5). Participants with left heart disease or left heart failure were excluded (WHO Group 2). Participants could be receiving prostacyclin or sildenafil therapy at baseline, and participants who previously discontinued either bosentan, sitaxsentan, or both, due to liver function test abnormalities were eligible.

ELIGIBILITY:
Summarized Inclusion Criteria:

1. 18 years of age or older
2. Current diagnosis of PH associated with an acceptable etiology as outlined in the protocol, including: PH due to the following etiologies: 1) PAH including idiopathic and familial PAH and PAH associated with collagen vascular disease, congenital systemic-to-pulmonary shunts (including Eisenmenger's syndrome), human immunodeficiency virus (HIV) infection, drugs and toxins, thyroid disorders, glycogen storage disease, Gaucher disease, hemoglobinopathies, and splenectomy (WHO Group 1); 2) PH associated with lung diseases and/or hypoxemia, including chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), sleep-disordered breathing, and alveolar hypoventilation disorders (WHO Group 3); 3) PH due to proximal or distal chronic thromboembolic obstruction (WHO Group 4); and 4) PH due to sarcoidosis (WHO Group 5).
3. Stable regimen (within four weeks) of chronic prostanoid, PDE-5 inhibitor, calcium channel blocker, or 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor therapy
4. Right heart catheterization completed prior to screening must meet pre-specified criteria
5. Female participants of childbearing potential must have a negative serum pregnancy test and must agree to use a reliable double method of contraception until study completion and for at least four weeks following their final study visit.
6. Male participants must be informed of the potential risks of testicular tubular atrophy and infertility associated with taking ambrisentan and queried regarding his understanding of the potential risks as described in the Informed Consent Form.

Summarized Exclusion Criteria:

1. Participation in a previous clinical study with ambrisentan
2. Bosentan or sitaxsentan use within four weeks prior to the screening visit
3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) lab value that is greater than 3 times the upper limit of normal at the screening visit
4. Pulmonary function tests not meeting the following pre-specified criteria: 1) mean pulmonary arterial pressure (PAP) >= 25 mm Hg; 2) PVR > 3 mm Hg/L/min; 3) pulmonary capillary wedge pressure (PCWP) or left ventricle end diastolic pressure (LVEDP) < 15 mm Hg; 4) total lung capacity (TLC) >= 70% of predicted normal for participants without ILD or >= 60% of predicted normal in participants with ILD; forced expiratory volume in 1 second (FEV1) >= 65% of predicted normal in participants without COPD or >= 50% of predicted normal in participants with COPD
5. Contraindication to treatment with endothelin receptor antagonist (ERA)
6. History of malignancies other than basal cell carcinoma of the skin or in situ carcinoma of the cervix within the past five years
7. Female participant who is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J Rubin, MD, Principal Investigator — University of California, San Diego
Locations (39):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Ltd, Phoenix, Arizona
  - UCSD Medical Center, Thornton Hospital, La Jolla, California
  - Greater Los Angeles, VA Medical Center, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Pulmonary Hypertension Clinic Mount Sinai Medical Center, Miami Beach, Florida
  - Suncoast Lung Center, Sarasota, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Atlanta Institute for Medical Research, Inc., Decatur, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Adult Congenital Heart Service, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Medicine & Dentistry of New Jersey, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Presbyterian Pulmonary Hypertension Center, New York, New York
  - Mary Parkes Asthma Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Legacy Clinical Northwest, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lexington Pulmonary and Critical Care, Lexington, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia Health Sciences Center, Charlottesville, Virginia
- Australia (2):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Royal Perth Hospital, Perth
- Canada (3):
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- See also: Related Info — http://www.gilead.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between September 2006 and January 2008 and the study was conducted between August 2006 and May 2009 in 39 centers in the United States, Australia and Canada
Pre-assignment Details: The screening period was 4 weeks. Participants who received bosentan or sitaxsentan within 4 weeks prior to the screening visit were excluded.
Groups:
- Ambrisentan: Eligible participants received 5 mg ambrisentan once daily for the first 24 weeks. One dose reduction to 2.5 mg was permitted during the 24-week fixed-dose treatment period if the participant did not tolerate the study drug. After the initial 24-week treatment period, investigators could adjust the study drug dose as clinically indicated (available doses were 2.5, 5, and 10 mg).
Period: Overall Study
Arm/Group | Ambrisentan
Started | 224
Completed | 155
Not Completed | 69
Not completed — Adverse Event | 40
Not completed — Withdrawal by Subject | 10
Not completed — Not compliant | 6
Not completed — Lost to Follow-up | 1
Not completed — Addition of other PAH therapeutic agent | 1
Not completed — Lung transplant | 3
Not completed — Physician Decision | 2
Not completed — Partipant moved away | 1
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in 6 Minute Walk Distance (6MWD)
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Last Observation Carried forward. 4 participants were excluded from the analysis due to lack of post-baseline 6MWD data.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 220
meters | 20.5 (65.64) [21 to 48]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test on change from Baseline to Week 24; Mean Difference (Net) = 20.5, 95% CI [11.8 to 29.3], Standard Deviation 65.64

2. Secondary Outcome: Change From Baseline to Week 24 in Borg Dyspnea Index
Description: Change from Baseline to Week 24 in Borg Dyspnea Index. The Borg Dyspnea Index of Perceived Exertion Scores range from 0 to 10. Best and Worst values are: 0 (Best) to 10 (Worst). Scales are described as rating of breathlessness and its description: 0= none; 0.5= very,very slight (just noticeable); 1= very slight; 2=slight; 3= moderate; 4= somewhat severe; 5= severe; 6 (in between severe and very severe); 7= very severe; 8 (in between very, very severe and maximum); 9= very, very severe; and 10= maximum.
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Last Observation Carried forward. 4 participants were excluded from the analysis due to lack of post-baseline Borg Dyspnea Index data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 220
Units on a scale | -0.5 (2.18) [-0.8 to -0.3]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test on change from Baseline to Week 24; Mean Difference (Net) = -0.5, 95% CI [-0.8 to -0.3], Standard Deviation 2.11

3. Secondary Outcome: Change From Baseline to Week 48 in Borg Dyspnea Index
Description: Change from Baseline to Week 48 in Borg Dyspnea Index. The Borg Dyspnea Index of Perceived Exertion Scores range from 0 to 10. Best and Worst values are: 0 (Best) to 10 (Worst). Scales are described as rating of breathlessness and its description: 0= none; 0.5= very,very slight (just noticeable); 1= very slight; 2=slight; 3= moderate; 4= somewhat severe; 5= severe; 6 (in between severe and very severe); 7= very severe; 8 (in between very, very severe and maximum); 9= very, very severe; and 10= maximum.
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Observed data. 114 participants were excluded from the analysis due to lack of Week 48 Borg Dyspnea Index data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 110
Units on a scale | -0.6 (1.91) [-1.0 to -0.2]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Paired t-test on change from Baseline to Week 48; Mean Difference (Net) = -0.6, 95% CI [-1.0 to -0.2]

4. Secondary Outcome: Percent Change From Baseline to Week 24 in B-type Natriuretic Peptide (BNP)
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Last Observation Carried forward. 10 participants were excluded from the analysis due to lack of baseline or post-baseline BNP data.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change in BNP
Arm/Group | Ambrisentan
Number analyzed (Participants) | 214
Percent change in BNP | -25.5 [-33.6 to -16.3]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; Percent change from baseline = -25.5, 95% CI [-33.6 to -16.3] — Percent change from baseline derived from Geometric Mean Ratio

5. Secondary Outcome: Percent Change From Baseline to Week 48 in BNP
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Observed data. 111 participants were excluded from the analysis due to lack of baseline or Week 48 BNP data.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change in BNP
Arm/Group | Ambrisentan
Number analyzed (Participants) | 112
Percent change in BNP | -29.2 [-39.8 to -16.6]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; Percent change from baseline = -29.2, 95% CI [-39.8 to -16.6] — Percent change from baseline derived from Geometric Mean Ratio

6. Secondary Outcome: Change From Baseline to Week 24 in WHO Functional Class
Description: Change from baseline in World Health Organization functional class (WHO) at Week 24 is the incidence of participants that improved, had no change, or worsened. WHO categories are 1 to 4 with the worse category at 4. Improvement = a category change from baseline of <= -1: change of -3 (eg, WHO from 4 to 1), change of -2 (eg, WHO from 3 to 1), change of -1 (eg, WHO from 2 to 1). Inversely, participants worsening are those with a category change from baseline of at least +1. No change in WHO functional class represents the percentage of participants with a change in category from baseline of 0.
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Last Observation Carried Forward. 3 participants were not analyzed due to lack of post-baseline WHO functional class data.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 221
Percentage of participants
  -3 | 0
  -2 | 0.9
  -1 | 22.2
  0 | 70.1
  1 | 6.8
  2 | 0
  3 | 0
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — Statistical test performed on actual change from baseline WHO functional Class (eg, a change from WHO Class III to II is -1; a change from WHO Class IV to II is -2; etc)

7. Secondary Outcome: Change From Baseline to Week 48 in WHO Functional Class
Description: Change from baseline in WHO at Week 48 is expressed as the incidence of participants that improved, had no change or worsened. WHO categories range from 1 to 4 with the worse category at 4. Improvement = a category change from baseline of <= -1: change of -3 (eg, WHO from 4 to 1), change of -2 (eg, WHO from 3 to 1), change of -1 (eg, WHO from 2 to 1). Inversely, participants worsening are those with a category change from baseline of at least +1. No change in WHO functional class represents the percentage of participants with a change in category from baseline of 0.
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Observed Data. 3 participants were not analyzed due to lack of post-baseline WHO functional class data.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 119
Percentage of participants
  -3 | 0
  -2 | 1.7
  -1 | 34.5
  0 | 57.1
  1 | 6.7
  2 | 0
  3 | 0
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Change From Baseline to Week 24 in SF-36 Health Survey Physical Functioning Scale
Description: Change from baseline to Week 24 in the SF-36 health survey physical functioning scale. 10 activities rated by health limitations using 3 categories (1= Yes, limited a lot; 2= Yes, limited a little; and 3= No, not limited at all). The best score is 3 and the worst score is 1. Scores are transformed by subtracting the unit by the lowest raw score and dividing by the raw score range. The scores are then standardized with the 1998 General United States (US) population mean and standard deviation (SD). Finally, the scores are transformed to the norm-based scoring with a mean of 50 and SD of 10.
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Last Observation Carried forward. 26 participants were excluded from the analysis due to lack of baseline or post-baseline SF-36 data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 198
Units on a scale | 2.88 (7.943) [-29.5 to 25.3]
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test on change from Baseline to Week 24

9. Secondary Outcome: Change From Baseline to Week 48 in SF-36 Health Survey Physical Functioning Scale
Description: Change from baseline to Week 48 in the SF-36 health survey physical functioning scale. 10 activities are rated by health limitations using 3 categories (1= Yes, limited a lot; 2= Yes, limited a little; and 3= No, not limited at all). The best score is 3 and the worst score is 1. Scores are transformed by subtracting the unit by the lowest raw score and dividing by the raw score range. The scores are then standardized with the 1998 General US population mean and standard deviation. Finally, the scores are transformed to the norm-based scoring with a mean of 50 and standard deviation of 10.
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Last Observation Carried forward. 25 participants were excluded from the analysis due to lack of baseline or post-baseline SF-36 data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ambrisentan
Number analyzed (Participants) | 199
Units on a scale | 2.80 (8.634)
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Paired t-test on change from Baseline to Week 48

10. Secondary Outcome: Percent of Participants With no Clinical Worsening of Pulmonary Hypertension (PH) at Week 24
Description: Clinical worsening: occurrence of death, lung transplantation, hospitalization for PH, atrial septostomy, a change to chronic prostanoid or sildenafil treatment due to protocol-defined worsening criteria, or study withdrawal due to the addition of other clinically approved PH therapeutic agents
Time Frame: Baseline to Week 24
Population: Full analysis set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 89.4
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 89.4, 95% CI [84.4 to 92.8] — Estimate obtained through Kaplan-Meier methods

11. Secondary Outcome: Percent of Participants With no Clinical Worsening of PH at Week 48
Description: as for outcome 10
Time Frame: Baseline to Week 48
Population: Full analysis set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 84.1
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 84.1, 95% CI [78.2 to 88.6] — Estimate obtained through Kaplan-Meier methods

12. Secondary Outcome: Failure-free Treatment Status
Description: Defined by occurrence of death, lung transplantation, or study withdrawal due to the addition of other clinically approved PAH therapeutic agents
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 95.3
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 95.3, 95% CI [91.4 to 97.4] — Estimate obtained through Kaplan-Meier methods

13. Secondary Outcome: Failure-free Treatment Status
Description: as for outcome 12
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 92.9
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 92.9, 95% CI [88.3 to 95.8] — Estimate obtained through Kaplan-Meier methods

14. Secondary Outcome: Monotherapy Treatment Status
Description: Defined by no addition of sildenafil, iloprost, treprostinil, or epoprostenol to ongoing ambrisentan treatment
Time Frame: Baseline to Week 24
Population: Full Analysis Set - Subset of participants who were not receiving other PH therapy at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 107
Percentage of participants | 95.0
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 95.0, 95% CI [88.5 to 97.9] — Estimate obtained through Kaplan-Meier methods

15. Secondary Outcome: Monotherapy Treatment Status
Description: Defined by no addition of sildenafil, iloprost, treprostinil, or epoprostenol to ongoing ambrisentan treatment
Time Frame: Baseline to Week 48
Population: Full Analysis Set - Subset of participants who were not receiving other PH therapy at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 107
Percentage of participants | 90.0
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 90.0, 95% CI [81.6 to 94.7] — Estimate obtained through Kaplan-Meier methods

16. Secondary Outcome: Long-term Survival
Description: Defined as not dying during study participation
Time Frame: Baseline to Week 24
Population: Full Analysis Set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 97.1
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 97.1, 95% CI [93.6 to 98.7] — Estimate obtained through Kaplan-Meier methods

17. Secondary Outcome: Long-term Survival
Description: Defined as not dying during study participation
Time Frame: Baseline to Week 48
Population: Full Analysis Set. Participants who were lost to follow-up were censored at the date of last contact.
Measure: Number; unit: Percentage of participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 224
Percentage of participants | 95.3
Statistical Analysis 1: Comparison: Ambrisentan; Test type: Superiority or Other; percent event free = 95.3, 95% CI [91.2 to 97.6] — Estimate obtained through Kaplan-Meier methods

ADVERSE EVENTS:
Time Frame: AEs were to be collected during study and up to 72 hours after last dose. SAEs, including deaths, that occurred during the study or within 4 weeks of receiving the last dose of study drug, whether or not related to study drug, were to be reported.
Arm/Group | Ambrisentan
Serious Adverse Events (participants affected / at risk) | 97/224
Other Adverse Events (participants affected / at risk) | 203/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=224)
alanine aminotransferase increased (Investigations) | 2
aspartate aminotransferase increased (Investigations) | 2
drug interaction (General disorders) | 1
international normalised ratio increased (Investigations) | 3
muscle tightness (Musculoskeletal and connective tissue disorders) | 1
narcotic intoxication (Injury, poisoning and procedural complications) | 1
neutropenia (Blood and lymphatic system disorders) | 1
abdominal pain (Gastrointestinal disorders) | 3
abscess limb (Infections and infestations) | 2
atrial fibrillation (Cardiac disorders) | 3
atrial flutter (Cardiac disorders) | 2
atrioventricular block third degree (Cardiac disorders) | 1
autoimmune hepatitis (Hepatobiliary disorders) | 1
blood glucose increased (Investigations) | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
bronchiectasis (Infections and infestations) | 1
bronchitis (Infections and infestations) | 2
bronchitis acute (Infections and infestations) | 1
cardiac failure congestive (Cardiac disorders) | 2
cardio-respiratory arrest (Cardiac disorders) | 2
cellulitis (Infections and infestations) | 2
central line infection (Infections and infestations) | 1
cerebrovascular accident (Nervous system disorders) | 2
chest pain (General disorders) | 5
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7
deep vein thrombosis (Vascular disorders) | 1
dehydration (Metabolism and nutrition disorders) | 1
device related infection (Infections and infestations) | 1
diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
dizziness (Nervous system disorders) | 3
drug hypersensitivity (General disorders) | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
endocarditis (Infections and infestations) | 1
enteritis infectious (Infections and infestations) | 1
enterobacter infection (Infections and infestations) | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
face oedema (General disorders) | 1
femur fracture (Injury, poisoning and procedural complications) | 1
fluid overload (Metabolism and nutrition disorders) | 2
gastroenteritis viral (Infections and infestations) | 1
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
headache (Nervous system disorders) | 1
hypervolaemia (Metabolism and nutrition disorders) | 1
hypoglycaemia (Metabolism and nutrition disorders) | 1
hypokalaemia (Metabolism and nutrition disorders) | 3
hyponatraemia (Metabolism and nutrition disorders) | 2
hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
influenza (Infections and infestations) | 1
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
left ventricular failure (Cardiac disorders) | 1
liver function test abnormal (Investigations) | 3
lower respiratory tract infection (Infections and infestations) | 2
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
mental status changes (Psychiatric disorders) | 1
migraine (Nervous system disorders) | 1
migraine with aura (Nervous system disorders) | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 1
non-cardiac chest pain (General disorders) | 1
oedema (General disorders) | 1
oedema peripheral (General disorders) | 3
ovarian cyst ruptured (Reproductive system and breast disorders) | 1
pericardial effusion (Cardiac disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
pneumonia (Infections and infestations) | 15
pneumonia bacterial (Infections and infestations) | 1
productive cough (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 8
pulomonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
raynaud's phenomenon (Vascular disorders) | 1
recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
renal failure (Renal and urinary disorders) | 1
renal failure acute (Renal and urinary disorders) | 2
renal impairment (Renal and urinary disorders) | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
respiratory tract infection (Infections and infestations) | 2
right ventricular failure (Cardiac disorders) | 16
sedation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
sepsis (Infections and infestations) | 4
shock haemorrhagic (Vascular disorders) | 1
sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1
spinal compression fracture (Injury, poisoning and procedural complications) | 1
syncope (Nervous system disorders) | 1
systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
transaminase increased (Investigations) | 2
transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
tremor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
urinary retention (Renal and urinary disorders) | 1
urinary tract infection (Infections and infestations) | 2
vaginal haemorrhage (Reproductive system and breast disorders) | 1
anaemia (Blood and lymphatic system disorders) | 1
iron deficiency anaemia (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
cardiac arrest (Cardiac disorders) | 1
cardiac failure (Cardiac disorders) | 1
cor pulmonale (Cardiac disorders) | 2
palpitations (Cardiac disorders) | 1
supraventricular tachycardia (Cardiac disorders) | 1
diverticular perforation (Gastrointestinal disorders) | 1
gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
peritonitis (Gastrointestinal disorders) | 1
appendicitis (Infections and infestations) | 2
arthritis infective (Infections and infestations) | 1
catheter sepsis (Infections and infestations) | 1
gastroenteritis (Infections and infestations) | 1
sepsis syndrome (Infections and infestations) | 1
septic shock (Infections and infestations) | 1
upper respiratory tract infection (Infections and infestations) | 2
accidental overdose (Injury, poisoning and procedural complications) | 2
fall (Injury, poisoning and procedural complications) | 1
fibula fracture (Injury, poisoning and procedural complications) | 1
thrombosis in device (Injury, poisoning and procedural complications) | 1
tibia fracture (Injury, poisoning and procedural complications) | 1
hepatic enzyme increased (Investigations) | 1
diabetes mellitus (Metabolism and nutrition disorders) | 1
hyperkalaemia (Metabolism and nutrition disorders) | 3
fracture nonunion (Musculoskeletal and connective tissue disorders) | 1
scleroderma (Musculoskeletal and connective tissue disorders) | 1
presyncope (Nervous system disorders) | 1
subarachnoid haemorrhage (Nervous system disorders) | 1
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
anxiety (Psychiatric disorders) | 1
confusional state (Psychiatric disorders) | 1
depression (Psychiatric disorders) | 1
nervousness (Psychiatric disorders) | 1
panic attack (Psychiatric disorders) | 1
suicidal ideation (Psychiatric disorders) | 1
suicide attempt (Psychiatric disorders) | 1
nephrolithiasis (Renal and urinary disorders) | 1
renal failure chronic (Renal and urinary disorders) | 1
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
skin ulcer (Skin and subcutaneous tissue disorders) | 1
hypotension (Vascular disorders) | 1
vasculitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=224)
arthralgia (Musculoskeletal and connective tissue disorders) | 20
back pain (Musculoskeletal and connective tissue disorders) | 24
brain natriuretic peptide increased (Investigations) | 18
cough (Respiratory, thoracic and mediastinal disorders) | 29
depression (Psychiatric disorders) | 27
diarrhoea (Gastrointestinal disorders) | 22
dizziness (Nervous system disorders) | 30
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48
fatigue (General disorders) | 39
flushing (Vascular disorders) | 16
headache (Nervous system disorders) | 63
hypokalemia (Metabolism and nutrition disorders) | 19
insomnia (Psychiatric disorders) | 17
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 41
nausea (Gastrointestinal disorders) | 33
oedema peripheral (General disorders) | 95
pain in extremity (Musculoskeletal and connective tissue disorders) | 24
upper respiratory tract infection (Infections and infestations) | 54
urinary tract infection (Infections and infestations) | 22
vomiting (Gastrointestinal disorders) | 18
anaemia (Blood and lymphatic system disorders) | 17
palpitations (Cardiac disorders) | 17
abdominal pain (Gastrointestinal disorders) | 12
constipation (Gastrointestinal disorders) | 19
chest pain (General disorders) | 16
pyrexia (General disorders) | 12
bronchitis (Infections and infestations) | 17
nasopharyngitis (Infections and infestations) | 12
sinusitis (Infections and infestations) | 17
international normalised ratio increased (Investigations) | 15
fluid overload (Metabolism and nutrition disorders) | 12
anxiety (Psychiatric disorders) | 12
epistaxis (Respiratory, thoracic and mediastinal disorders) | 16
rash (Skin and subcutaneous tissue disorders) | 13
hypotension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs have right disclose data upon publication of a multi-center publication coordinated by Sponsor or 18 months after Study is completed at all sites if multi-center publication is not submitted by Sponsor within 12 mos. PI to furnish Sponsor with copy of proposed disclosure at least 90 days prior to proposed disclosure. Sponsor has right to ensure accuracy of disclosure and request deletion of confidential information. Sponsor may not make editorial changes to the results or conclusions.